CLINICAL TRIAL: NCT04101292
Title: Endoscopic Optical Imaging for Precision Oncology Treatment Applied to Colorectal Tumours
Brief Title: Endoscopic Optical Imaging for Precision Oncology Treatment Applied to Colorectal Tumours (Elios-Color-on-Specimen)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with the provision of equipment encountered during the study could not be resolved, making it impossible to take the images planned for the main objective of the study.
Sponsor: IHU Strasbourg (Other)
Collaborators: ARC Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-004
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: Fluorescence; Antibody; Bevacizumab; IRDye800; Hyperspectral imaging; Light-CT Scanner; Tumour detection; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescence characterization (Experimental)
  Interventions: Other: Characterization of tumor tissue by fluorescence

INTERVENTIONS:
Other: Characterization of tumor tissue by fluorescence — * HSI Imaging of the resected specimen, from the serum and the mucous side
  * FF-OCT imaging of the tumor and the healthy tissue biopsies
  * Local application of Bevacizumab-IRDye800CW and visualization with the Surgvision Explorer system
  * Standard anti-VEGF Immunohistochemistry and pathology

SUMMARY:
The Institute of Image-Guided Surgery (IHU) of Strasbourg is a translational research Institute aiming to develop hybrid surgery techniques. The IHU-SPECTRA research unit, entirely dedicated to the development of fluorescence-guided surgery, was set up to test several innovations as part of a large-scale project (ELIOS: Endoscopic Luminescent Imaging for Precision Oncology Surgery), funded by the ARC Foundation for Cancer Research. The proposed research protocol is part of the ELIOS project and targets in particular colon tumours.

The Holy Grail in oncology surgery is the radical removal of cancer cells in order to reduce the rate of tumour recurrences and increase the tumour's free survival.

The administration of a tumour-specific antibody, which fluoresces in the Near-Infrared ranges and which could be univocally recognized at a tumour cellular level, could provide a rapid and accurate evaluation of radical tumour removal.

The University Medical Center Groningen (UMCG) has developed a fluorescent tracer coupling Bevacizumab (which targets the Vascular Endothelial Growth Factor = VEGF) with a fluorescent dye, the IRDye800. The initial human results are very promising and no adverse events linked to the fluorescent molecule have been reported.

In parallel, an alternative optical technique that does not require the use of a fluorophore, the Hyperspectral Imaging (HSI), is a relatively new method used in image-guided and precision surgery. The company Diaspective Vision GmbH (Pepelw, Germany) produces a HSI camera, the TIVITA system, enabling to obtain spectral information from the tissues. The main advantage of HSI over fluorescence imaging is in that it is a contrast-free imaging and intrinsically quantitative although it does not provide real-time videos.

Another innovative optical imaging technology available at the IHU is FF-OCT (Light-CT Scanner, LLTechSAS, Paris, France) which allows non-destructive and high-resolution optical biopsy without tissue treatment.

The working hypothesis is that molecular fluorescence enhanced-reality allows greater precision in the differentiation of tumour tissue and healthy tissue in patients with colorectal cancer compared to the immunohistochemistry conventionally used in anatomopathology.

In parallel, this technique will be compared to hyperspectral imaging (HSI TIVITA system) and optical imaging (FF-OCT system), two potentially advantageous methods for the detection of tumour tissue.

DETAILED DESCRIPTION:
The Institute of Image-Guided Surgery (IHU) of Strasbourg is a translational research Institute aiming to develop hybrid surgery techniques, less invasive and image-guided to improve the therapeutic results, in the emerging context of the precision medicine.

One of those expanding technique is fluorescence imaging that can guide the surgical procedure very accurately.

The IHU-SPECTRA research unit, entirely dedicated to the development of fluorescence-guided surgery, was set up at the IHU Strasbourg. Currently represented by a network of scientists from different fields and by industrial and academic partners in France and abroad, its short-term goals are mainly the implementation and evaluation in current clinical practice of the techniques already developed. In the long term, it is planned to test several innovations as part of a large-scale project (ELIOS: Endoscopic Luminescent Imaging for Precision Oncology Surgery), funded by the ARC Foundation for Cancer Research.

The proposed research protocol is part of the ELIOS project and targets in particular colon tumours.

The Holy Grail in oncology surgery is the radical removal of cancer cells in order to reduce the rate of tumour recurrences and increase the tumour's free survival. Tumour involvement at the resection margins is the most important predictor of tumour recurrence, leading to high recurrence rate.

However, surgery and other minimally-invasive ablative procedures are currently limited by 1) the need of wide removal of healthy tissue in order to ensure negative margins (which might lead to functional deficits and increases the risks of complications) and 2) frozen sections analysis to verify the surgical margins. They are time consuming and require considerable human resources.

The administration of a tumour-specific antibody, which fluoresces in the Near-Infrared ranges and which could be univocally recognized at a tumour cellular level, could provide a rapid and accurate evaluation of radical tumour removal. In the context of precision surgery, the development of tumour-specific fluorescent probes has made remarkable advances over recent years, with promising pre-clinical proofs of the concept, allowing for the enhanced identification of tumour residuals and metastatic lymph nodes. Recently, in a pioneer paper published on Nature, the first human case of tumour-specific fluorescence-guided surgery has been reported. Authors could remove effectively 34 intra-peritoneal implants of ovarian cancer metastasis, which were completely invisible at the naked eye. This impressive proof of the concept highlights clearly the potential impact of intraoperative tumour-specific molecular fluorescence imaging.

There is an increasing number of targeted probes which are being developed to visualize cancer cells, enabling early stage cancer detection and precise tumour resection. Particularly interesting is the strategy of coupling a fluorescent dye (IRDye800CW) with the humanized monoclonal antibodies, currently used in anticancer therapy.

The University Medical Center Groningen (UMCG), which is a strong partner of the IHU-SPECTRA unit, has developed a fluorescent tracer coupling Bevacizumab (which targets the Vascular Endothelial Growth Factor = VEGF) with the IRDye800.

The initial human results obtained together with the company Surgvision (Groningue, Pays-Bas) are very promising and have reported no adverse events linked to the fluorescent.

Bevacizumab-IRDye800CW can be either intravenously perfused or locally applied, the local application being more efficient than the perfusion.

In parallel, an alternative optical technique that does not require the use of a fluorophore will be tested. This technology, the Hyperspectral Imaging (HSI), is a relatively new method used in image-guided and precision surgery, which has shown promising results for recognition/characterization of tissues/tumours, and comprehensive assessment of physiologic tissue parameters, such as perfusion, oxygenation, and water content. Hence, it has been applied predominantly in wound imaging and -management in plastic surgery transplants, vascular surgery, chronical wounds and burn injuries.

The HSI system from a German start-up (Diaspective Vision GmbH, Pepelw, Germany) has been acquired. The company produces a HSI camera, the TIVITA system, enabling to obtain spectral information from the tissues. The only limitation, when applied to minimally-invasive surgery, is in that the TIVITA provides pictures and not real-time videos.

The main advantage of HSI over fluorescence imaging is in that it is a contrast-free imaging and intrinsically quantitative. Those characteristics make of the HSI a very promising tool in image-guided surgery, and open several windows of opportunity in terms of research programs towards miniaturization and optimization of the image-flow and artificial intelligence (AI) algorithms of tissue recognition.

Another innovative optical imaging technology available at the IHU is FF-OCT (Light-CT Scanner, LLTechSAS, Paris, France). This technology allows non-destructive and high-resolution optical biopsy without tissue treatment. The images are generated by measuring the backscattered light produced by the interaction between light and tissues of different indices. This technology has already shown its significant potential in oncology, particularly for ovarian, brain, mammary and pancreatic tissues. If validated, it could in the future complement or even replace traditional pathology, since it provides high-resolution images in a short time, without the need for treatment or staining.

The working hypothesis is that molecular fluorescence enhanced-reality allows greater precision in the differentiation of tumour tissue and healthy tissue in patients with colorectal cancer compared to the immunohistochemistry conventionally used in anatomopathology.

In parallel, this technique will be compared to hyperspectral imaging (HSI TIVITA system) and optical imaging (FF-OCT system), two potentially more advantageous methods for the detection of tumour tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman over 18 years old
2. Patient with colorectal cancer
3. Patient able to receive and understand information related to the study and to give written informed consent.
4. Patient affiliated to the French social security system

Exclusion Criteria:

1. Pregnant or lactating patient
2. Patient in exclusion period (determined by a previous or a current study)
3. Patient under guardianship or trusteeship
4. Patient under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the sensitivity of Bevacizumab-IRDye800 to visualize tumour tissue relative to surrounding healthy tissue by the means of fluorescence intensity measurements | 1 day
  Correlation between the fluorescence signal intensity of Bevacizumab-IRDye800CW emitted by tumours and sensed by near-infrared imaging systems compared to the fluorescence emitted by healthy tissue
Evaluation of the sensitivity of Bevacizumab-IRDye800 to visualize tumour tissue compared to anti-VEGF antibodies by the means of fluorescence intensity measurements | 1 day
  Correlation between the fluorescence signal intensity of Bevacizumab-IRDye800CW emitted by tumours and sensed by near-infrared imaging systems compared to VEGF expression levels in immunohistochemistry and histological diagnosis

SECONDARY OUTCOMES:
Ability of Hyperspectral Imaging (HSI) to detect the tumour area on the serosal side before marking the margins of resection by the means of spectral signature characterization | 1 day
  Correlation of the spectral signatures between healthy and tumour bearing segments from the serosa side, obtained by HSI before marking the margins of resection
Ability of HSI to detect the tumour area on the serosal side after marking the margins of resection by the means of spectral signature characterization | 1 day
  Correlation of the spectral signatures between healthy and tumour bearing segments from the serosa side, obtained by HSI after marking the margins of resection
Ability of HSI to determine the tumour stage from the serosal side | 1 day
  Correlation of the tumour stage specific spectral features obtained from the serosal side with the final histopathological tumour stage
HSI's ability to identify the tumoural and healthy tissue from the mucosal side compared to the results provided by histopathology and immunohistochemistry (IHC). | 1 day
  Determination of the presence or absence of spectral signature obtained by HSI on two regions of interest (one located in the tumour and the other outside the tumour) and correlation with standard pathology and IHC
Level of accuracy of resection of a fluorescence-guided tumour determined by the presence or absence of tumourous cells on resection margins by histological examination | 1 day
  Evaluation of the efficiency of fluorescence-guided full-thickness resection by histopathologically evaluating the presence or absence of tumours on resection margins
Level of accuracy of fluorescence microscopy compared to ImmunoHistoChemistry | 1 day
  Comparison of the fluorescence signal intensity detected within and outside the tumour by fluorescence microscopy and immunohistochemical analysis
Level of accuracy of Full-field optical coherence tomography (FF-OCT) by the means of a qualitative analysis | 1 day
  Qualitative analysis with FF-OCT of untreated biopsies compared to frozen sections and standard pathology

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg; Michele DIANA, MD, Study Director — IHU Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harlaar NJ, Koller M, de Jongh SJ, van Leeuwen BL, Hemmer PH, Kruijff S, van Ginkel RJ, Been LB, de Jong JS, Kats-Ugurlu G, Linssen MD, Jorritsma-Smit A, van Oosten M, Nagengast WB, Ntziachristos V, van Dam GM. Molecular fluorescence-guided surgery of peritoneal carcinomatosis of colorectal origin: a single-centre feasibility study. Lancet Gastroenterol Hepatol. 2016 Dec;1(4):283-290. doi: 10.1016/S2468-1253(16)30082-6. Epub 2016 Sep 17. PMID 28404198
- [Background] Diana M. Enabling precision digestive surgery with fluorescence imaging. Transl Gastroenterol Hepatol. 2017 Nov 21;2:97. doi: 10.21037/tgh.2017.11.06. eCollection 2017. No abstract available. PMID 29264435
- [Background] Lamberts LE, Koch M, de Jong JS, Adams ALL, Glatz J, Kranendonk MEG, Terwisscha van Scheltinga AGT, Jansen L, de Vries J, Lub-de Hooge MN, Schroder CP, Jorritsma-Smit A, Linssen MD, de Boer E, van der Vegt B, Nagengast WB, Elias SG, Oliveira S, Witkamp AJ, Mali WPTM, Van der Wall E, van Diest PJ, de Vries EGE, Ntziachristos V, van Dam GM. Tumor-Specific Uptake of Fluorescent Bevacizumab-IRDye800CW Microdosing in Patients with Primary Breast Cancer: A Phase I Feasibility Study. Clin Cancer Res. 2017 Jun 1;23(11):2730-2741. doi: 10.1158/1078-0432.CCR-16-0437. Epub 2016 Nov 9. PMID 28119364
- [Background] Tjalma JJ, Garcia-Allende PB, Hartmans E, Terwisscha van Scheltinga AG, Boersma-van Ek W, Glatz J, Koch M, van Herwaarden YJ, Bisseling TM, Nagtegaal ID, Timmer-Bosscha H, Koornstra JJ, Karrenbeld A, Kleibeuker JH, van Dam GM, Ntziachristos V, Nagengast WB. Molecular Fluorescence Endoscopy Targeting Vascular Endothelial Growth Factor A for Improved Colorectal Polyp Detection. J Nucl Med. 2016 Mar;57(3):480-5. doi: 10.2967/jnumed.115.166975. Epub 2015 Dec 17. PMID 26678613
- [Background] Rosenthal EL, Warram JM, de Boer E, Basilion JP, Biel MA, Bogyo M, Bouvet M, Brigman BE, Colson YL, DeMeester SR, Gurtner GC, Ishizawa T, Jacobs PM, Keereweer S, Liao JC, Nguyen QT, Olson JM, Paulsen KD, Rieves D, Sumer BD, Tweedle MF, Vahrmeijer AL, Weichert JP, Wilson BC, Zenn MR, Zinn KR, van Dam GM. Successful Translation of Fluorescence Navigation During Oncologic Surgery: A Consensus Report. J Nucl Med. 2016 Jan;57(1):144-50. doi: 10.2967/jnumed.115.158915. Epub 2015 Oct 8. PMID 26449839
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Kellokumpu I, Vironen J, Kairaluoma M, Jantunen I, Kautiainen H, Nuorva K. Quality of surgical care, local recurrence, and survival in patients with low- and midrectal cancers following multimodal therapy. Int J Colorectal Dis. 2012 Jan;27(1):111-20. doi: 10.1007/s00384-011-1322-5. Epub 2011 Oct 26. PMID 22038306
- [Background] Metildi CA, Felsen CN, Savariar EN, Nguyen QT, Kaushal S, Hoffman RM, Tsien RY, Bouvet M. Ratiometric activatable cell-penetrating peptides label pancreatic cancer, enabling fluorescence-guided surgery, which reduces metastases and recurrence in orthotopic mouse models. Ann Surg Oncol. 2015;22(6):2082-7. doi: 10.1245/s10434-014-4144-1. Epub 2014 Oct 16. PMID 25319581
- [Background] Metildi CA, Kaushal S, Luiken GA, Hoffman RM, Bouvet M. Advantages of fluorescence-guided laparoscopic surgery of pancreatic cancer labeled with fluorescent anti-carcinoembryonic antigen antibodies in an orthotopic mouse model. J Am Coll Surg. 2014 Jul;219(1):132-41. doi: 10.1016/j.jamcollsurg.2014.02.021. Epub 2014 Mar 2. PMID 24768506
- [Background] Metildi CA, Kaushal S, Pu M, Messer KA, Luiken GA, Moossa AR, Hoffman RM, Bouvet M. Fluorescence-guided surgery with a fluorophore-conjugated antibody to carcinoembryonic antigen (CEA), that highlights the tumor, improves surgical resection and increases survival in orthotopic mouse models of human pancreatic cancer. Ann Surg Oncol. 2014 Apr;21(4):1405-11. doi: 10.1245/s10434-014-3495-y. Epub 2014 Feb 6. PMID 24499827
- [Background] Metildi CA, Tang CM, Kaushal S, Leonard SY, Magistri P, Tran Cao HS, Hoffman RM, Bouvet M, Sicklick JK. In vivo fluorescence imaging of gastrointestinal stromal tumors using fluorophore-conjugated anti-KIT antibody. Ann Surg Oncol. 2013 Dec;20 Suppl 3(0 3):S693-700. doi: 10.1245/s10434-013-3172-6. Epub 2013 Aug 14. PMID 23943029
- [Background] Tran Cao HS, Kaushal S, Metildi CA, Menen RS, Lee C, Snyder CS, Messer K, Pu M, Luiken GA, Talamini MA, Hoffman RM, Bouvet M. Tumor-specific fluorescence antibody imaging enables accurate staging laparoscopy in an orthotopic model of pancreatic cancer. Hepatogastroenterology. 2012 Sep;59(118):1994-9. doi: 10.5754/hge11836. PMID 22369743
- [Background] van Dam GM, Themelis G, Crane LM, Harlaar NJ, Pleijhuis RG, Kelder W, Sarantopoulos A, de Jong JS, Arts HJ, van der Zee AG, Bart J, Low PS, Ntziachristos V. Intraoperative tumor-specific fluorescence imaging in ovarian cancer by folate receptor-alpha targeting: first in-human results. Nat Med. 2011 Sep 18;17(10):1315-9. doi: 10.1038/nm.2472. PMID 21926976
- [Background] McElroy M, Kaushal S, Luiken GA, Talamini MA, Moossa AR, Hoffman RM, Bouvet M. Imaging of primary and metastatic pancreatic cancer using a fluorophore-conjugated anti-CA19-9 antibody for surgical navigation. World J Surg. 2008 Jun;32(6):1057-66. doi: 10.1007/s00268-007-9452-1. PMID 18264829
- [Background] Hall MA, Pinkston KL, Wilganowski N, Robinson H, Ghosh P, Azhdarinia A, Vazquez-Arreguin K, Kolonin AM, Harvey BR, Sevick-Muraca EM. Comparison of mAbs targeting epithelial cell adhesion molecule for the detection of prostate cancer lymph node metastases with multimodal contrast agents: quantitative small-animal PET/CT and NIRF. J Nucl Med. 2012 Sep;53(9):1427-37. doi: 10.2967/jnumed.112.106302. Epub 2012 Aug 7. PMID 22872743
- [Background] Nakajima T, Mitsunaga M, Bander NH, Heston WD, Choyke PL, Kobayashi H. Targeted, activatable, in vivo fluorescence imaging of prostate-specific membrane antigen (PSMA) positive tumors using the quenched humanized J591 antibody-indocyanine green (ICG) conjugate. Bioconjug Chem. 2011 Aug 17;22(8):1700-5. doi: 10.1021/bc2002715. Epub 2011 Jul 27. PMID 21740058
- [Background] Rosbach KJ, Williams MD, Gillenwater AM, Richards-Kortum RR. Optical molecular imaging of multiple biomarkers of epithelial neoplasia: epidermal growth factor receptor expression and metabolic activity in oral mucosa. Transl Oncol. 2012 Jun;5(3):160-71. doi: 10.1593/tlo.11310. Epub 2012 Jun 1. PMID 22741035
- [Background] Nagengast WB, Hartmans E, Garcia-Allende PB, Peters FTM, Linssen MD, Koch M, Koller M, Tjalma JJJ, Karrenbeld A, Jorritsma-Smit A, Kleibeuker JH, van Dam GM, Ntziachristos V. Near-infrared fluorescence molecular endoscopy detects dysplastic oesophageal lesions using topical and systemic tracer of vascular endothelial growth factor A. Gut. 2019 Jan;68(1):7-10. doi: 10.1136/gutjnl-2017-314953. Epub 2017 Dec 15. No abstract available. PMID 29247063
- [Background] Hartmans E, Tjalma JJJ, Linssen MD, Allende PBG, Koller M, Jorritsma-Smit A, Nery MESO, Elias SG, Karrenbeld A, de Vries EGE, Kleibeuker JH, van Dam GM, Robinson DJ, Ntziachristos V, Nagengast WB. Potential Red-Flag Identification of Colorectal Adenomas with Wide-Field Fluorescence Molecular Endoscopy. Theranostics. 2018 Feb 5;8(6):1458-1467. doi: 10.7150/thno.22033. eCollection 2018. PMID 29556334
- [Background] Peters IT, Stegehuis PL, Peek R, Boer FL, van Zwet EW, Eggermont J, Westphal JR, Kuppen PJ, Trimbos JB, Hilders CG, Lelieveldt BP, van de Velde CJ, Bosse T, Dijkstra J, Vahrmeijer AL. Noninvasive Detection of Metastases and Follicle Density in Ovarian Tissue Using Full-Field Optical Coherence Tomography. Clin Cancer Res. 2016 Nov 15;22(22):5506-5513. doi: 10.1158/1078-0432.CCR-16-0288. Epub 2016 May 16. PMID 27185369
- [Background] Binding J, Ben Arous J, Leger JF, Gigan S, Boccara C, Bourdieu L. Brain refractive index measured in vivo with high-NA defocus-corrected full-field OCT and consequences for two-photon microscopy. Opt Express. 2011 Mar 14;19(6):4833-47. doi: 10.1364/OE.19.004833. PMID 21445119
- [Background] Assayag O, Antoine M, Sigal-Zafrani B, Riben M, Harms F, Burcheri A, Grieve K, Dalimier E, Le Conte de Poly B, Boccara C. Large field, high resolution full-field optical coherence tomography: a pre-clinical study of human breast tissue and cancer assessment. Technol Cancer Res Treat. 2014 Oct;13(5):455-68. doi: 10.7785/tcrtexpress.2013.600254. Epub 2013 Aug 31. PMID 24000981
- [Background] van Manen L, Stegehuis PL, Farina-Sarasqueta A, de Haan LM, Eggermont J, Bonsing BA, Morreau H, Lelieveldt BPF, van de Velde CJH, Vahrmeijer AL, Dijkstra J, Mieog JSD. Validation of full-field optical coherence tomography in distinguishing malignant and benign tissue in resected pancreatic cancer specimens. PLoS One. 2017 Apr 17;12(4):e0175862. doi: 10.1371/journal.pone.0175862. eCollection 2017. PMID 28414765